CLINICAL TRIAL: NCT04419337
Title: Comparison of Combined Pioglitazone and SGLT2 Inhibitors vs. DPP4 Inhibitors in Diabetic Patients With Ischemic Stroke: Rationale and Study Design
Brief Title: Pioglitazone and SGLT2 Inhibitors vs. DPP4 Inhibitors in Patients With Stroke
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Collaborators: National Taiwan University Hospital (Other); Chiayi Christian Hospital (Other); Tainan Sin-lau Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MOST 108-2314-B-182-017-
Record Dates: First submitted 2020-02-26; First posted 2020-06-05 (Actual); Last update posted 2023-03-30 (Actual); Status verified 2023-03

CONDITIONS: Diabetes Mellitus; Stroke
Keywords: stroke; diabetes mellitus; sodium-glucose transport protein 2 inhibitor; pioglitazone
MeSH Terms: conditions — Diabetes Mellitus; Stroke | interventions — Metformin; Pioglitazone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active arm (Experimental): metformin+pioglitazone+an SGLT2 inhibitor
  Interventions: Drug: Metformin plus Pioglitazone plus an SGLT2 inhibitor
- Control arm (Active Comparator): metformin + DPP4 inhibitors
  Interventions: Drug: Metformin plus Pioglitazone plus an SGLT2 inhibitor

INTERVENTIONS:
Drug: Metformin plus Pioglitazone plus an SGLT2 inhibitor — Patients assigned to active group will stop their prior oral antidiabetic drugs and receive combination of metformin, pioglitazone, and an SGLT2 inhibitor (empagliflozin or dapagliflozin or canagliflozin) and dose will be adjusted by their physicians.

SUMMARY:
Introduction: An optimal combination of antidiabetic drugs for diabetic patients with ischemic stroke is not well-established. The objective of this randomized trial is to evaluate whether combination of pioglitazone and a sodium glucose cotransporter 2 (SGLT-2) inhibitor, compared with a dipeptidyl peptidase-4 (DPP-4) inhibitor, reduces recurrent stroke in diabetic patients with recent ischemic stroke.

Methods and analysis: The trial is a randomized, parallel-group study conducted at 7 hospitals in Taiwan. Inclusion criteria are adult patients with a history of ischemic stroke within 3 months, diabetes mellitus with Hba1C > 7%, taking metformin currently or previously, and estimated glomerular filtration rate ≥ 45 mL/min/1.73 m2. Eligible patients who sign the informed consent forms will be randomly assigned in a 1:1 ratio to receive either combination of pioglitazone and an SGLT2 inhibitor (empagliflozin or dapagliflozin or canagliflozin) vs. a DPP4 inhibitor. Primary outcome is change in HbA1C between 6 months and baseline in active vs comparator groups. Additional biomarker outcomes are change in hs-CRP insulin resistance, B type natriuretic peptide, and urine albumin creatinine ratio between 6 months and baseline.

Ethics and dissemination Study protocol was approved by the Institutional Review Board of Chang Gung Memorial Hospital, Chiayi Branch, Taiwan (201702353A3, 201802340A3 and 201902176A3). All participants will be required to sign and date an informed consent form. Study findings will be disseminated via a peer-reviewed journal.

ELIGIBILITY:
Inclusion Criteria:

1. Ischemic stroke within 3 months of randomization
2. Type 2 diabetes mellitus and Hba1C > 7.0% and under metformin therapy currently or previously
3. Estimated glomerular filtration rate (eGFR) ≥ 45 mL/min/1.73 m2
4. Age ≥ 20 y at study entry
5. Ability and willingness to provide informed consent

Exclusion Criteria:

1. History of congestive heart failure (NYHA class 1-4)
2. History of bladder cancer
3. History of repeated (> 2 episodes) urinary tract infection or genital tract infection
4. Irreversible medical conditions with predicted survival < 1 years
5. Current use of an insulin
6. Current use of a glucagon-like peptide-1 receptor agonist
7. Current use of pioglitazone or an SGLT-2 inhibitor

Ages: 20 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-09-15 (Actual); Primary Completion 2023-07-31 (Estimated); Study Completion 2024-01-31 (Estimated)

PRIMARY OUTCOMES:
HbA1C | 6 months from baseline in active vs control arms
  blood test to evaluate glycemic control

SECONDARY OUTCOMES:
UACR | 6 months from randomization in active vs control arms
  to evaluate microalbuminuria
hs-CRP | 6 months from randomization
  to evaluate hs-CRP in active vs control arms
NT-proBNP | 6 months from randomization
  to evaluate NT-proBNP in active vs control arms
insulin resistance | 6 months from randomization
  Insulin resistance will be evaluated by Homeostatic Model Assessment for Insulin Resistance (HOMA-IR)

CONTACTS AND LOCATIONS:
Overall Officials: Meng Lee, MD, Principal Investigator — Chang Gung Memorial Hospital, Chiayi Branch
Locations (1):
- Chang Gung Memorial Hospital, Chiayi Branch, Chiayi City, Taiwan

IPD SHARING:
Plan to Share IPD: No